CLINICAL TRIAL: NCT03041246
Title: The Influence of Manual Fascial Manipulation on the Function of the Pelvic Floor in Pregnant Women
Brief Title: Manual Fascial Manipulation in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3722-16-SMC
Record Dates: First submitted 2017-01-24; First posted 2017-02-02 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: On enrollment, dividing the healthy ( n=40) from the pathological function of the pelvic floor ( n=40). From the second group, randomizing the groups to study group: recieving pelvic floor fascial mobilization (PFFM) treatment (n=20)compared to control group (n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group - Treatment with PFFM (Experimental): Manual treatment for the pelvic floor will be provided in two sessions two weeks apart as long as guidance towards exercise for strengthening of the pelvic floor
  Interventions: Procedure: Pelvic floor fascial mobilization
- Control group - (No Intervention): Guidance towards exercise for strengthening of the pelvic floor with no other interventional treatment.

INTERVENTIONS:
Procedure: Pelvic floor fascial mobilization — The manual manipulation of the pelvic floor involves intra vaginal superficial as well as pelvic skin area pressure points.
  Arms: Study group - Treatment with PFFM

SUMMARY:
Pregnancy and vaginal delivery are considered as the main risk factors for damage to the pelvic floor. There are various ways to measure the strength of the pelvic floor and to evaluate functional problems. Manual mobilization of the pelvic floor is a well-known treatment modality, however, ample knowledge exists on the efficacy of physiotherapy and exercise for improvement of pelvic floor function and strength. The aim of this study is to analyze the influence of pelvic floor fascial mobilization (PFFM) technique on the function and strength of the pelvic floor muscles as well as parameters presumed to be influenced by the strength of the pelvic floor in pregnant women.

DETAILED DESCRIPTION:
Pregnancy and vaginal delivery are considered as the main risk factors for damage to the pelvic floor at various degrees, starting at mild stress incontinence and up to fool fecal incontinence as well as pelvic pains or urination difficulties.

There are various ways to measure the strength of the pelvic floor and to evaluate functional problems. Measured the strength of the pelvic floor muscles by physical examination according to Oxford Grading Scale (scale of 0-5) as well as by using Perineometer device, were equally efficient and well correlated. Other modalities such as the use of surface electro myography (EMG), that presents the level of the muscle electrical activity and expiration volumes and the strength of the pelvic floor muscles were also positively correlated to the strength of the pelvic floor. Recent studies presented dysfunction of pelvic floor during pregnancy as well as in the postpartum period by the use of pelvic floor disability index 20 (PFDI20) questionnaire validated in Hebrew.

Ample knowledge exists on the efficacy of physiotherapy and exercise for improvement of pelvic floor function and strength, however, prolonged and continuous exercise is needed to achieve good results as well as compliance and perseverance. The long-term effect is unwieldly.

Manual mobilization of the pelvic floor is a well-known treatment modality. However the literature regarding the effect of this technique is sparse. A recent series of case reports presented immediate and major improvement of pelvic floor dysfunction after manual mobilization. The peripartum period is critical for the function of the pelvic floor however the yield of manual therapy on function and strength of the pelvic floor was not evaluated in pregnant women. We hypothesize that manual therapy can improve the strength and the function of the pelvic floor within a short time span and this can be objectively measured by common and well used parameters The aim of this study is to analyze the influence of pelvic floor fascial mobilization (PFFM) on the function and strength of the pelvic floor muscles as well as parameters presumed to be influenced by the strength of the pelvic floor in pregnant women

Materials and methods

The study will involve number of phases:

Phase one: Screening and enrollment of patients Women followed at the high risk pregnancy clinic at the Sheba medical center, who carry singleton pregnancy at the ages of 20-45 years old and about to have their 2nd to 4th delivery (primiparous and multiparous women) will be examined for the following parameters: demographic and medical data, focused interview for symptoms of pelvic floor dysfunction including urination and fecal function as well as pelvic floor pain, manual assessment according the Oxford grading scale will be performed, and the strength of the pelvic floor measured by the use of Perineometer (Peritron 'AV' Combined Anal & Vaginal Perineometer NEW MODEL). Other parameters that will be measured include: mobilization of the pelvic-femoral joint, Forced expiratory volume 1 (FEV1) (a connection was shown between FEV1, intraabdominal pressure and the strength of the pelvic floor, assessment of vocal quality ( analyzed by communication clinician, repeat assessment will be performed after two weeks and after 4 weeks, estimated assessment time - 20 Min) 80 women are expected to be enrolled.

Phase Two Women who will fulfill one or more of the following parameters will be enrolled to the second phase of the study . (n=40)

1. Oxford grading scale ≤3/5
2. Pelvic floor strength assessed by perineometer≤ 30 cm/h20
3. Clinical symptoms of urine, flatus or fecal incontinence
4. Pelvic floor, hip joint or pelvic joints pain

Randomization will be performed to one of two groups:

Group A-Control group (n=20) Group B-Study group (n=20) Guidance towards exercise for strengthening of the pelvic floor will be provided for both groups. Study group will be treated manually for the pelvic floor in two sessions two weeks apart. The manual manipulation of the pelvic floor will involve intra vaginal superficial as well as pelvic skin area pressure points. The manipulation will not involve the cervix uterus or rectum. Each session will lasts one hour

Both groups will be assessed by ultrasound for blood flow in the middle cerebral artery, umbilical artery and uterine artery as part of the parameters that may show benefit to the fetus due to pelvic floor mobilization.

Reassessment of all the women and repeat treatment for the study group will be performed after two and four weeks from the primary assessment.

The study will be performed at a high risk pregnancy clinic at the Sheba medical center. Women will be enrolled voluntarily with no financial benefit.

ELIGIBILITY:
Inclusion criteria:

1. Age 20-45 years old
2. Gestational age 24-30 weeks gestation
3. Singleton pregnancy
4. Expected second-4ourth delivery

Exclusion criteria

1. First delivery
2. Gestational age at more than 30 weeks gestation at enrollment
3. Premature contractions
4. Cervical insufficiency
5. Placenta previa
6. Placenta accrete
7. Multifetal pregnancy
8. Maternal chronic illness including connective tissue disease, neurological illness

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women that are pregnant
Enrollment: 80 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Contraction strength | Change of contraction strength is assessed - from baseline to 2 weeks after last treatment ( up to maximum of 1 month )
  Contraction strength assessed by Oxford grading scale
Contraction pressure | Change of contraction pressure is assessed - from baseline to 2 weeks after last treatment ( up to maximum of 1 month )
  Contraction pressure measured by using Peritron perineometer

SECONDARY OUTCOMES:
Symptoms associated with pelvic dysfunction | Change of pelvic dysfunction is assessed - from baseline to 2 weeks after last treatment ( up to maximum of 1 month )
  Assessment of symptoms associated with pelvic dysfunction: urinary incontinence, fecal incontinence, frequency and urgency (by the use of pelvic floor disability index 20 - a questionaire including 20 questions on pelvic floor function)
FEV1 | Change of FEV1 is assessed - from baseline to 2 weeks after last treatment ( up to maximum of 1 month )
  Forced expiratory volume 1
Voice Handicap Index - 10 among Hebrew speakers (VHI-10-HEB) questionaire | Change of VHI-10-HEB is assessed - from baseline to 2 weeks after last treatment ( up to maximum of 1 month )
  Evaluation of the validity of the voice handicap index that includes ten questions concerning voice usage among hebrew speakers

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batista EM, Conde DM, Do Amaral WN, Martinez EZ. Comparison of pelvic floor muscle strength between women undergoing vaginal delivery, cesarean section, and nulliparae using a perineometer and digital palpation. Gynecol Endocrinol. 2011 Nov;27(11):910-4. doi: 10.3109/09513590.2011.569603. Epub 2011 Apr 18. PMID 21500994
- [Background] Hallock JL, Handa VL. The Epidemiology of Pelvic Floor Disorders and Childbirth: An Update. Obstet Gynecol Clin North Am. 2016 Mar;43(1):1-13. doi: 10.1016/j.ogc.2015.10.008. PMID 26880504
- [Background] Navot S, Kalichman L. Hip and groin pain in a cyclist resolved after performing a pelvic floor fascial mobilization. J Bodyw Mov Ther. 2016 Jul;20(3):604-9. doi: 10.1016/j.jbmt.2016.04.005. Epub 2016 Apr 7. PMID 27634085
- [Background] Okido MM, Valeri FL, Martins WP, Ferreira CH, Duarte G, Cavalli RC. Assessment of foetal wellbeing in pregnant women subjected to pelvic floor muscle training: a controlled randomised study. Int Urogynecol J. 2015 Oct;26(10):1475-81. doi: 10.1007/s00192-015-2719-4. Epub 2015 Aug 21. PMID 26294205
- [Background] Petricelli CD, Resende AP, Elito Junior J, Araujo Junior E, Alexandre SM, Zanetti MR, Nakamura MU. Distensibility and strength of the pelvic floor muscles of women in the third trimester of pregnancy. Biomed Res Int. 2014;2014:437867. doi: 10.1155/2014/437867. Epub 2014 Apr 28. PMID 24877094
- [Background] Talasz H, Kofler M, Kalchschmid E, Pretterklieber M, Lechleitner M. Breathing with the pelvic floor? Correlation of pelvic floor muscle function and expiratory flows in healthy young nulliparous women. Int Urogynecol J. 2010 Apr;21(4):475-81. doi: 10.1007/s00192-009-1060-1. Epub 2009 Dec 8. PMID 19997721
- [Background] van Veelen GA, Schweitzer KJ, van der Vaart CH. Ultrasound imaging of the pelvic floor: changes in anatomy during and after first pregnancy. Ultrasound Obstet Gynecol. 2014 Oct;44(4):476-80. doi: 10.1002/uog.13301. PMID 24436146
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735